CLINICAL TRIAL: NCT05948878
Title: An Innovative Taping Technique for Improved Intravenous (IV) Catheter Securement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Pete Kovatsis, Principle Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-P00043126
Record Dates: First submitted 2022-11-28; First posted 2023-07-17 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Dislodged Catheter; Catheter Related Complication
Keywords: Catheter Taping Methods; Catheter securement; Catheters; Intravenous catheters

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrograde Directional Test (Active Comparator): Subjects during the Retrograde Directional Test will have the three taping methods placed on their left and/or right antecubital fossa region to superficially secure an IV catheter (i.e., the catheter will be placed on top of the participant's skin and not in the vein but will be taped as if the catheter was placed intravenously). Six total measurements will be obtained of which three will be using the Retrograde Directional Test (i.e., each taping method will undergo testing for each directional method). The order of placing the different taping methods and the direction testing will be randomized.
  Interventions: Device: Novel Taping Method; Device: BCH Emergency Department Taping Method; Device: Chevron Taping Method
- 90 Degrees Directional Test (Active Comparator): Subjects during the 90 Degrees Directional Test will have the three taping methods placed on their left and right antecubital fossa region, superficially taping an IV catheter (i.e., the catheter will be placed on top of the participant's skin and not in the vein but will be taped as if the catheter was placed intravenously). Six total measurements will be obtained of which three will be using the 90 Degrees Directional Test (i.e., each taping method will undergo testing for each directional method). The order of placing the different taping methods and the direction testing will be randomized.
  Interventions: Device: Novel Taping Method; Device: BCH Emergency Department Taping Method; Device: Chevron Taping Method

INTERVENTIONS:
Device: Novel Taping Method — Subjects will be asked to have the novel taping method placed on their left and right antecubital fossa region, superficially taping an IV catheter.
Device: BCH Emergency Department Taping Method — Subjects will be asked to have the BCH emergency department taping method placed on their left and right antecubital fossa region, superficially taping an IV catheter.
Device: Chevron Taping Method — Subjects will be asked to have the Chevron taping method placed on their left and right antecubital fossa region, superficially taping an IV catheter.

SUMMARY:
This is a prospective, single-blinded, randomized study to assess the ability of taping methods used to secure intravenous (IV) catheters to resist the IV from being pulled away from the skin. Participants will have IV catheters taped on top of the skin (without insertion into the skin) using three taping methods, BCH Emergency Department (BCH ED), Chevron, and our novel method. Six measurements will be obtained per subject (3 random taping methods measuring their resistance to force in two directions, retrograde direction or towards the wrist and 90-degree angle to the arm).

DETAILED DESCRIPTION:
Accidental removal of IV catheters delay patient care and can cause additional medical anxiety and pain that is heightened in the pediatric population. Moreover, such failed catheters create an increased burden economically and emotionally to patients, hospitals, and clinicians. To facilitate the most accurate, consistent results, a calibrated hand wheel test stand with a force gauge will be used to obtain force measurements. We will obtain the amount of force is required to remove the IV catheter form the skin of the subjects to compare the three taping measurements in two different directions. The retrograde direction will be pulling the IV distally from the IV site, towards the participant's wrist. The 90-degree angle will be pulling the IV medially away from the IV site.

ELIGIBILITY:
Inclusion Criteria:

* Employees of Boston Children's Hospital

Exclusion Criteria:

* Individuals under the direct supervision of any study investigators
* Individuals with excessive hair in/near the antecubital fossa region on either arm
* Individuals with fragile and/or non-intact skin in/near the antecubital fossa region
* Individuals who have adhesive allergies
* Individuals who have already participated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
The Force (Newtons) Required to Dislodge an IV Catheter Secured by the Chevron, BCH ED, and Novel Taping Methods Using a Force Gauge in the retrograde direction. | Until the tape is dislodged- approximately 15 seconds
  We will examine the maximum force the Chevron, BCH ED, and Novel taping methods can withstand as measured by the force gauge in the retrograde direction, distally from the insertion site.
The Force (Newtons) Required to Dislodge an IV Catheter Secured by the Chevron, BCH ED, and Novel Taping Methods Using a Force Gauge in a 90 degrees direction. | Until the tape is dislodged- approximately 15 seconds
  We will examine the maximum force the Chevron, BCH ED, and Novel taping methods can withstand as measured by the force gauge in a 90 degrees direction, medially from the insertion site.

CONTACTS AND LOCATIONS:
Overall Officials: Pete Kovatsis, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No